CLINICAL TRIAL: NCT01169909
Title: The Use of Ranibizumab to Control Pterygium Growth in Recurrences and in Non-surgical Primary Lesions.
Brief Title: Efficacy and Safety of Sub-tenon Ranibizumab for Recurrent Pterygia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Linda Rose, Principal Investigator, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-117
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Pterygium
Keywords: Pterygium
MeSH Terms: conditions — Pterygium | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab treatment (Experimental): Patients will receive a sub-tenons injection of Ranibizumab 0.5mg, to be repeated twice with 30 day intervals between each dose.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Subtenon injections of Ranibizumab 0.5mg will be given, and repeated twice with 30 day intervals between each dose. Note, after an amendment in February 2011, this dose was increased to 2mg with the same schedule.

SUMMARY:
Ranibizumab, an effective antineovascular drug, will be studied for safety and efficacy in pterygium, a neovascular disorder of the ocular surface.

DETAILED DESCRIPTION:
Ptergyia are chronic fibrovascular lesions of the ocular surface. This study is designed to look for a signal of efficacy when the lesions are in a phase of active vascular growth. This phase is most often caught in a newly recurring pterygia post-operatively.

Patients identified with actively growing lesions, will be offered local injections directly beneath the lesions. They will be examined for any adverse side effects and regression of the lesion.

ELIGIBILITY:
Inclusion Criteria:

Patients with actively growing pterygia, either surgical recurrences, or non-surgical primary lesions.

Exclusion Criteria:

* Pregnancy
* History of CVA
* Monocular patients
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety | Within the first 30 days after injection
  The following safety criteria will be monitored: subjective complaints, objective signs of inflammation, intraocular pressure, tear film and ocular surface integrity.

SECONDARY OUTCOMES:
Regression of pterygium | Within 30 days after drug injection
  Regression of the lesion will be determined by measurement if the horizontal extension of the lesion relative to the limbus, and by photographic comparison incorporating software analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Health Science Center, Albuquerque, New Mexico, United States